CLINICAL TRIAL: NCT06174766
Title: A Multicenter, Randomized, Double-blind, Phase 3 Study to Evaluate Efficacy and Safety of HGP2102 in Patients With Essential Hypertension
Brief Title: A Study to Evaluate Efficacy and Safety of HGP2102 in Essential Hypertension Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-ENCORE-301
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental1 (Experimental): Take HGP2102-1 once daily for 4 weeks orally, and then take HGP2102-2 once daily for 6 weeks orally.
  Interventions: Drug: HGP2102-1; Drug: HGP2102-2
- Experimental2 (Experimental): Take HGP2102-1 once daily for 10 weeks orally.
  Interventions: Drug: HGP2102-1
- Active Comparator (Active Comparator): Take RLD2209-1 once daily for 4 weeks orally, and then take RLD2209-2 once daily for 6 weeks orally.
  Interventions: Drug: RLD2209-1; Drug: RLD2209-2

INTERVENTIONS:
Drug: HGP2102-1 — Test drug
  Arms: Experimental1; Experimental2
Drug: HGP2102-2 — Test drug
  Arms: Experimental1
Drug: RLD2209-1 — Control drug
  Arms: Active Comparator
Drug: RLD2209-2 — Control drug
  Arms: Active Comparator

SUMMARY:
A Multicenter, Randomized, Double-blind, Phase 3 Study to Evaluate the Efficacy and Safety of HGP2102 in patients with Essential Hypertension

ELIGIBILITY:
Inclusion Criteria:

1. Subjects whose clinic blood pressure measured in visit 1 corresponds to the following conditions

   * sitSBP<180 mmHg and sitDBP<110mg for patients receiving any BP-lowering drug within 1 month prior to Visit 1
   * 140mmHG≤sitSBP<180mmHg and 60mmHg≤sitDBP<110mmHg
2. Subjects whose clinic and ambulatory blood pressure measured in visit 2 corresponds to the following conditions

   * 24h-ABPM: 130mmHg≤ SBP <170mmHg
   * clinic BP: 140 mmHg ≤ sitSBP < 180 mmHg and 60 mmHg ≤ sitDBP < 110 mmHg

Exclusion Criteria:

1. Difference between arms greater than 20 mmHg for mean sitSBP or 10mmHg for mean sitDBP at Visit 1
2. Patients who have taken more than three components of Blood pressure medication within 3 months prior to Visit 1
3. Orthostatic hypotension with symptoms within 3 months prior to visit 1
4. Secondary hypertension patient or suspected to be
5. Uncontrolled type II diabetes mellitus (HbA1c > 9%) or type I diabetes mellitus
6. Severe heart disease or severe neurovascular disease
7. Moderate or malignant retinopathy
8. Severe renal diseases (eGFR<30mL/min/1.73m2)
9. Severe or active hepatopathy (AST or ALT ≥ 2 times of normal range)
10. Hypokalemia or Hyperkalemia (K<3.5mmol/L or K ≥ 5.5mmol/L)
11. Hyponatremia or Hypernatremia (Na<135mmol/L or Na ≥ 155mmol/L)
12. History of malignancy tumor
13. History of alcohol or drug abuse
14. Positive to pregnancy test, nursing mother, intention on pregnancy
15. Considered by investigator as not appropriate to participate in the clinical study with other reason

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 24 hours ambulatory systolic blood pressure | baseline, 10 weeks

SECONDARY OUTCOMES:
Change from baseline in 24 hours ambulatory systolic blood pressure | baseline, 4 weeks
Change from baseline in 24 hours ambulatory diastolic blood pressure | baseline, 4 weeks, 10 weeks
Change from baseline in 24 hours ambulatory pulse pressure | baseline, 4 weeks, 10 weeks
Change from baseline in diurnal ambulatory systolic blood pressure | baseline, 4 weeks, 10 weeks
Change from baseline in diurnal ambulatory diastolic blood pressure | baseline, 4 weeks, 10 weeks
Change from baseline in diurnal ambulatory pulse pressure | baseline, 4 weeks, 10 weeks
Change from baseline in nocturnal ambulatory systolic blood pressure | baseline, 4 weeks, 10 weeks
Change from baseline in nocturnal ambulatory diastolic blood pressure | baseline, 4 weeks, 10 weeks
Change from baseline in nocturnal ambulatory pulse pressure | baseline, 4 weeks, 10 weeks
Change from baseline in sitting systolic blood pressure | baseline, 4 weeks, 10 weeks
Change from baseline in sitting diastolic blood pressure | baseline, 4 weeks, 10 weeks
Change from baseline in sitting pulse pressure | baseline, 4 weeks, 10 weeks
Proportion of subjects achieving blood pressure control | baseline, 4 weeks, 10 weeks
Blood pressure response rate | baseline, 4 weeks, 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sevrance hosptal, Seodaemun-gu, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No